CLINICAL TRIAL: NCT03306485
Title: Evaluation of Diagnostic Performances of Esophageal Post Prandial High Resolution Impedance- Manometry (HRIM) in Patients With Gastro-esophageal Reflux Disease (GERD) Resistant to Proton Pump Inhibitor (PPI) Treatment : Pilot Study (MHR POST-PRANDIALE)
Brief Title: Post Prandial High Resolution Impedance- Manometry
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0427
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Gastro-esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with GERD symptoms refractory to PPI therapy: Patients with proven GERD (gastro-esophageal reflux disease) off PPI (proton pump inhibitor) (Los Angeles grade B, C or D esophagitis and/or esophageal acid exposure > 5% on pH monitoring performed off PPI).
  These patients have persistent heartburn and/or regurgitation despite double dose proton pump inhibitor. Patients are referred for esophageal high resolution impedance manometry and ambulatory 24-h pH-impedance monitoring on proton pump inhibitor.
  Interventions: Other: Correlating the number of reflux episodes detected on 1-h post prandial esophageal high resolution manometry combined and those detected on ambulatory 24-h pH-impedance monitoring performed on PPI

INTERVENTIONS:
Other: Correlating the number of reflux episodes detected on 1-h post prandial esophageal high resolution manometry combined and those detected on ambulatory 24-h pH-impedance monitoring performed on PPI — Esophageal high resolution impedance manometry (HRIM) consists of introducing a transnasal probe to record esophageal contractility (manometry), bolus transit (impedance) but also the occurrence of reflux episodes. Ambulatory 24-h pH-impedance monitoring consists of recording the occurrence of reflux episodes by introducing a transnasal catheter into the esophagus. After inserting the transnasal HRIM probe and the pH-impedance catheter, both HRIM and 24-h pH-impedance recordings are started. The patient is instructed to eat a meal that induces reflux symptoms (the patient brings his own meal). One hour the end of the meal, the HRIM probe is removed. The patient is discharged at home and the 24-h pH-impedance monitoring is continued. The patient is coming back 24-h after catheter insertion to stop the pH-impedance recording and remove the catheter.

SUMMARY:
Nine to 30% of the population suffers from gastro-esophageal reflux disease (GERD) - suggestive symptoms (heartburn, regurgitation, chest pain, chronic couch, sore throat). Proton pump inhibitor (PPI) is usually the first line treatment. However 20 to 60% of patients have persistent symptoms on proton pump inhibitor. Complementary examinations are then required to determine the cause of persistent symptoms (non compliance to treatment, persistent esophageal acid exposure despite proton pump inhibitor, non acid reflux, reflux hypersensitivity, functional symptoms, rumination syndrome…). The gold standard to detect reflux episodes in patients on proton pump inhibitor therapy is 24-h ambulatory esophageal pH-impedance monitoring. Esophageal High Resolution Impedance-Manometry might help to determine gastro-esophageal reflux disease mechanisms especially when performed post prandially. Further some publications demonstrated that the number of reflux episodes detected during the post prandial period might be well correlated to the total number of reflux episodes recorded during 24 h.

The hypothesis of this study is that 1-hour post prandial esophageal High Resolution Impedance-Manometry might be useful to diagnose gastro-esophageal reflux disease and can replace in some instances 24-h esophageal pH-impedance monitoring. Therefore the aim is to compare the number of reflux episodes detected with esophageal High Resolution Impedance-Manometry performed during 1-h post prandial period to the total number of reflux episodes detected during 24-h ambulatory esophageal pH-impedance monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both gender older than 18 years
* Patient referred for post prandial esophageal high resolution manometry combined with impedance and ambulatory 24-h pH-impedance monitoring on proton pump inhibitor
* Heartburn and/or regurgitation despite double dose proton pump inhibitor therapy
* Proven Gastro-esophageal reflux disease off proton pump inhibitor (Los Angeles grade B, C or D esophagitis and/or esophageal acid exposure > 5% on esophageal pH monitoring off proton pump inhibitor)
* Absence of major esophageal motility disorders (achalasia, esophago-gastric junction outflow obstruction, esophageal spasm, jackhammer esophagus, absent contractions)
* Patient who does not decline to participate to the study

Exclusion Criteria:

* Patient younger than 18 years
* Pregnancy or breast feeding
* Previous history of esophago-gastric surgery ( including anti-reflux surgery, Heller myotomy, bariatric surgery)
* Patient with severe renal insufficiency
* Patient with severe cardiac insufficiency
* Patient legally incompetent or unable to give consent
* Patient who declines to participate to the study
* Participation to another study at the same time

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Gastro-esophageal reflux disease symptoms refractory to proton pump inhibitor therapy
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
High Resolution Impedance Manometry | 1 hour
  Number of reflux episodes detected on high resolution impedance manometry during the one hour following the meal
24-h pH-impedance | 24 hour
  Number of reflux episodes detected on 24-h ambulatory esophageal pH-impedance monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Exploration Fonctionnelle Digestive, Hôpital Edouard Herriot, Lyon, France, Lyon, France

IPD SHARING:
Plan to Share IPD: No